CLINICAL TRIAL: NCT02533557
Title: A Randomized Comparison Between 1 Plane-2 Injection and 2 Plane-2 Injection Ultrasound-guided Supraclavicular Brachial Plexus Block (US-SCBPB) in Upper Extremity Surgery
Brief Title: Comparison 1 Plane-2 Injection and 2 Plane-2 Injection Ultrasound-guided Supraclavicular Brachial Plexus Block
Acronym: US-SCBPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Mi Geum Lee, assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GBIRB2015-45
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Radius Fractures
Keywords: brachial plexus block; nerve stimulator; ultrasound
MeSH Terms: conditions — Radius Fractures | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2P2I group (Experimental): subcutaneous injection is done widely. A nerve stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) attached to a nerve stimulator (Stimuplex HNS12; B. Braun, Melsungen, Germany) is advanced via an ultrasound in-plane approach. After the needle is penetrated the nerve sheath with a direction of downward, the nerve stimulator is then turned on. If hand muscle twitching is observed even at 0.3 mA, LA 15 mL (lidocaine mixed with epinephrine) is injected. After that, the stimulating needle is re-advanced at the behind site of the initial puncture site. And the needle is penetrated the nerve sheath with a direction of upward, and then the same process is performed and LA 15 mL is injected.
  Interventions: Device: stimuplex insulated needle; Drug: lidocaine mixed with epinephrine
- 1P2I group (Active Comparator): subcutaneous injection is done widely. A nerve stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) attached to a nerve stimulator (Stimuplex HNS12; B. Braun, Melsungen, Germany) is advanced via an ultrasound in-plane approach. After the needle is penetrated the nerve sheath with a direction of downward, the nerve stimulator is then turned on. If hand muscle twitching is observed even at 0.3 mA, LA 15 mL (lidocaine mixed with epinephrine) is injected. After that, the stimulating needle is re-advanced with a direction of upward at the same puncture site and penetrated the nerve sheath. If hand muscle twitching is observed at 0.3 mA, LA 15 mL is injected.
  Interventions: Device: stimuplex insulated needle; Drug: lidocaine mixed with epinephrine

INTERVENTIONS:
Device: stimuplex insulated needle — 2P2I group: nerve stimulating needle is advanced twice with the up-down direction at the different puncture site and LA is injected 15 mL at a time.
  1P2I group: nerve stimulating needle is advanced twice with the up-down direction at the same puncture site and LA is injected 15 mL at a time.
  Other Names: D Plus B.Braun
Drug: lidocaine mixed with epinephrine — 2P2I group and 1P2I group use the same LA (1.5% lidocaine mixed with 1:200,000 epinephrine). But 2P2I group is injected LA at equally divided doses (15 mL at a time) with the up-down direction at the different puncture site. 1P2I group is injected LA at equally divided doses with the up-down direction at the same puncture site.
  Other Names: 1.5% lidocaine mixed with 1:200,000 epinephrine

SUMMARY:
The supraclavicular block can provide effective surgical anesthesia of the forearm and hand. There have been many different approaches to ultrasound-guided supraclavicular brachial plexus block (US-SCBPB) according to the needle injection site (e.g. corner pocket approach, cluster approach) or number of needling (single or double injection). Numerous studies demonstrates good results (e.g. faster onset time) when using double injections rather than single injection. But double injection does not guarantee complete sensory block because ulnar nerve tends to be spared by its anatomical location.

DETAILED DESCRIPTION:
The investigators hypothesized that double injection in different plane (we call this new approach as a 2 plane-2 injection approach;2P2I) would overcome the weakness of the existing double injection in same plane (we call this approach as a 1 plane-2 injection approach;1P2I) like "ulnar nerve sparing effect", and could have a good results (e.g. shortening the onset time or increasing rate of all four nerves block). Because 2P2I can achieve an effect of a "tridimensionally administered LA", rather 1P2I only achieve an effect of a " two-dimensionally administered LA".

ELIGIBILITY:
Inclusion Criteria:

* all patients anticipating surgery of the wrist or hand
* age: 18 to 80 years
* American Society of Anesthesiologists physical status (ASA): I or II

Exclusion Criteria:

* neuropathy in the operated limb
* ASA greater than III
* coagulation disorders
* known allergy to local anesthetics
* local infection at the puncture site
* chronic obstructive pulmonary disease or respiratory failure
* pregnancy or breast-feeding
* prior surgery in the supraclavicular region
* BMI ≥ 35 kg/㎡
* uncooperative patients
* patients' refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
rate of complete sensory blockade of all 4 nerves | check 30 minutes after performing the block at 5-minute intervals (from date of randomization until the date of first documented progression)
  If the sensory on the site under the control of all 4 (median, radial, ulnar, musculocutaneous) nerves is checked as 0 (just feeling of touch or none ) separately, it is considered as a complete sensory block.
  the investigators compare the rate of complete sensory block with 2P2I group and 1P2I group.

SECONDARY OUTCOMES:
the onset time | check 30 minutes after performing the block at 5-minute intervals(from date of randomization until the date of first documented progression)
  The investigators compare the onset time (time required to obtain of a sensory block at the surgical incision site) with 2P2I group and 1P2I group.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Geum Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Department of Anesthesiology and Pain Medicine, Gachon University Gil Medical Center, Incheon, Guwol-dong, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Techasuk W, Gonzalez AP, Bernucci F, Cupido T, Finlayson RJ, Tran DQ. A randomized comparison between double-injection and targeted intracluster-injection ultrasound-guided supraclavicular brachial plexus block. Anesth Analg. 2014 Jun;118(6):1363-9. doi: 10.1213/ANE.0000000000000224. PMID 24842181